CLINICAL TRIAL: NCT04334681
Title: Unroofing Curettage Versus Modified Limberg Flap in Pilonidal Disease: A Retrospective Cohort Study
Brief Title: Surgical Approach for Pilonidal Disease
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, principal investigator, Konya Meram State Hospital
Other Study IDs: pilonidal surgery group
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pilonidal Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UC Group: Patients operated on the un-roofing curettage method in the treatment of pilonidal disease will be analyzed in this group.
  Interventions: Procedure: Un-roofing curettage method
- LF Group: Patients who have been operated with the modified Limberg flap method after rhomboid excision in the treatment of pilonidal disease will be analyzed in this group.
  Interventions: Procedure: Modified Limberg Flap Group

INTERVENTIONS:
Procedure: Un-roofing curettage method — In this method, the roof of the pilonidal cyst is opened, and the inside is cleaned, and curettage is performed. The wound is closed with a dressing after hemostasis.
  Groups: UC Group
Procedure: Modified Limberg Flap Group — In this method, the pilonidal cyst is excised with a rhomboid incision and closed with the modified Limberg flap method.
  Groups: LF Group

SUMMARY:
In our hospital, between January 2013 and January 2017, those operated with the Modified Limberg flap method after the Rhomboid excision due to pilonidal disease, and those operated with the un-roofing curettage method will be screened retrospectively. Patients will be divided into two groups as Un-roofing curettage group (UC group) and the Modified Limberg Flap group (LF group). Operation time, hospital stay time, return to work time, recovery time, Time to walk without pain, days, Time to sit on the toilet without pain, days, Postoperative VAS and recurrence will be compared between both groups

DETAILED DESCRIPTION:
In our hospital, between January 2013 and January 2017, those operated with the Modified Limberg flap method after the Rhomboid excision due to pilonidal disease, and those operated with the un-roofing curettage method will be screened retrospectively. Patients who are well followed up will be included in the study. Demographic features will be recorded. Patients will be divided into two groups, the un-roofing curettage group (UC group) and the Modified Limberg Flap group (LF group). Surgery time, hospital stay, return to work time, recovery time, painless walking time, days, painless sitting time in the toilet, days, postoperative VAS, and recurrence will be compared between both groups. In addition, mobilization time, days, recovery time, days, exclusion time, days, wound infection, wound distribution will be compared between groups. The results will be analyzed with the SPSS statistics program. Factors affecting recurrence wound infection, recovery time, hospital stay, operation time, early mobilization will be evaluated by univariate and multivariate logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 70
* Patients with sufficient registration information
* Telephone-accessible patients

Exclusion Criteria:

* Patients under the age of 18
* Patients over 70 years old
* Common gluteal disease
* Diabetes mellitus
* Connective tissue disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Limberg flap after rhomboid excision and un-roofing curettage between January 2013 and January 2017 in our hospital constitute the study population.
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kemal Arslan, MD, Study Chair — Konya Research and Training Hospital
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mahdy T. Surgical treatment of the pilonidal disease: primary closure or flap reconstruction after excision. Dis Colon Rectum. 2008 Dec;51(12):1816-22. doi: 10.1007/s10350-008-9436-8. Epub 2008 Oct 21. PMID 18937009
- [Background] Kepenekci I, Demirkan A, Celasin H, Gecim IE. Unroofing and curettage for the treatment of acute and chronic pilonidal disease. World J Surg. 2010 Jan;34(1):153-7. doi: 10.1007/s00268-009-0245-6. PMID 19820992
- [Background] Karakayali F, Karagulle E, Karabulut Z, Oksuz E, Moray G, Haberal M. Unroofing and marsupialization vs. rhomboid excision and Limberg flap in pilonidal disease: a prospective, randomized, clinical trial. Dis Colon Rectum. 2009 Mar;52(3):496-502. doi: 10.1007/DCR.0b013e31819a3ec0. PMID 19333052
- [Result] Sahin A, Simsek G, Arslan K. Unroofing Curettage Versus Modified Limberg Flap in Pilonidal Disease: A Retrospective Cohort Study. Dis Colon Rectum. 2022 Oct 1;65(10):1241-1250. doi: 10.1097/DCR.0000000000002227. Epub 2022 May 24. PMID 34840296

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: When we planned to study, we estimated 200 patients. However, we reached 278 patient data and analyzed them.
Groups:
- LF Group: Patients who have been operated with the Limberg flap method after rhomboid excision in the treatment of pilonidal disease will be analyzed in this group.
  Limberg Flap Group: In this method, the pilonidal cyst is excised with a rhomboid incision and closed with the Limberg flap method.
Period: Overall Study
Arm/Group | UC Group | LF Group
Started | 135 | 143
Completed | 135 | 143
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UC Group | LF Group | Total
Number analyzed (Participants) | 135 | 143 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.35 (8.9) | 26.42 (7.9) | 25.90 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 115 | 127 | 242
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 135 | 143 | 278

OUTCOME MEASURES:

1. Primary Outcome: Mobilization Time,Days
Description: Time to return to the daily activities of the patients were measured.
Time Frame: 15 days
Measure: Median (Standard Deviation); unit: days
Groups:
- UC Group: Patients operated on the un-roofing curettage method in treating the pilonidal disease will be analyzed in this group.
  Un-roofing curettage method: In this method, the pilonidal cyst roof is opened, and the inside is cleaned, and curettage is performed. The wound is closed with a dressing after hemostasis.
- MLF Group: Patients who have been operated on with the modified Limberg flap method after rhomboid excision in the treatment of pilonidal disease will be analyzed in this group.
  Modified Limberg Flap Group: In this method, the pilonidal cyst is excised with a rhomboid incision and closed with the modified Limberg flap method.
Arm/Group | UC Group | MLF Group
Number analyzed (Participants) | 135 | 143
days | 3.21 (3.7) | 12.3 (7.3)

2. Primary Outcome: Number of Participants With Recurring Disease
Description: It has been reported in the literature that a five or ten year follow-up period is required for the effective evaluation of recurrence. In both groups, the number of recurrent patients during the follow-up period will be determined.
  Observation of the following findings on physical examination made a diagnosis of recurrence;
  * New sinus orifice formation,
  * Or discharge from the sinus orifice
Time Frame: Number of Participants with Recurring Disease, up to five years
Measure: Number; unit: participants
Arm/Group | MLF Group | UC Group
Number analyzed (Participants) | 143 | 135
participants | 6 | 2

3. Primary Outcome: Operation Time
Description: Mean operation time was determined in minutes in both groups.
Time Frame: operation time, up to 100 minutes
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | UC Group | MLF Group
Number analyzed (Participants) | 135 | 143
minute | 11.44 (3.56) | 52.47 (7.92)

4. Primary Outcome: Hospitalization Time
Description: In both groups, hospitalization will be determined as a day.
Time Frame: Hospitalization time, up to 15 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | UC Group | MLF Group
Number analyzed (Participants) | 135 | 143
days | 0.24 (0.45) | 1.07 (0.26)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | UC Group | LF Group
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/143
Serious Adverse Events (participants affected / at risk) | 1/135 | 2/143
Other Adverse Events (participants affected / at risk) | 2/135 | 12/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UC Group (N=135) | LF Group (N=143)
Hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Post-operative bleeding from the wound site
Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Postoperative hematoma (clotted blood accumulation) from the wound site
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UC Group (N=135) | LF Group (N=143)
Wound İnfection (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8) — wound infection development in the postoperative period
Wound dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) — wound dehiscence in the postoperative period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT04334681/Prot_SAP_001.pdf